CLINICAL TRIAL: NCT01302366
Title: A Phase II Trial of TBL12 Sea Cucumber Extract in Patients With Untreated Asymptomatic Myeloma
Brief Title: A Trial of TBL12 Sea Cucumber Extract in Patients With Untreated Asymptomatic Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to lack of funding
Sponsor: NYU Langone Health (Other)
Collaborators: Unicorn Pacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU# 10-02181
Record Dates: First submitted 2011-02-14; First posted 2011-02-24 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Myeloma
Keywords: multiple myeloma; myeloma; asymptomatic myeloma; smoldering myeloma; Asymptomatic (smoldering) myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sea cucumber extract (Experimental): TBL12 is administered orally at a dose of 2 units (of 20 mL each) twice a day, in 4-week cycles, until disease progression or there is sign of disease progression.
  Interventions: Drug: TBL12

INTERVENTIONS:
Drug: TBL12

SUMMARY:
This study proposes to determine the clinical activity of this agent in patients with asymptomatic multiple myeloma. It is believed that TBL12 will help delay the onset of active multiple myeloma, with very few-if any- side effects.

DETAILED DESCRIPTION:
Multiple myeloma is a cancer that evolves from a state known as Monoclonal Gammopathy of Undetermined Significance (MGUS), defined by parameters of M spike and bone marrow. After evolution to myeloma, patients may be asymptomatic, that is, without any endorgan disease of hypercalcemia, renal insufficiency, anemia or bone lesions. In asymptomatic myeloma (ASxM), there is no standard therapy. Thalidomide has been tried in patients with ASxM but with significant toxicity. The patients with ASxM are evaluable in terms of paraprotein measurements.

TBL12 sea cucumber extract has been shown to have a number of antitumor properties preclinically, including antiangiogenesis and direct tumor cytotoxicity. TBL12 has been used by a number of patients as a food supplement without any toxicity detected. The investigators thus propose to determine the clinical activity of this agent in patients with ASxM. Patients will be given TBL12 at the dose of 2 units of 20 mL each twice per day daily until disease progression and the effects on the paraprotein noted. Clinical effects seen will be correlated with any in vitro changes in angiogenesis in patient bone marrow samples. The results of this trial may form the basis for the use of this nontoxic agent in patients with the prodrome of or with other early cancers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based on standard criteria as follows:

Major Criteria

* Plasmacytomas on tissue biopsy
* Bone marrow plasmacytosis (> 30% plasma cells)
* Monoclonal immunoglobulin (Ig) spike on serum electrophoresis (IgG > 3.5 g/dL or IgA > 2.0 g/dL); kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis

Minor Criteria

* Bone marrow plasmacytosis (10 to 30% plasma cells)
* Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
* Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL

Any of the following sets of criteria will confirm the diagnosis of Multiple Myeloma:

* Any two of the major criteria
* Major criterion 1 plus minor criterion b, c
* Major criterion 3 plus minor criterion a or c
* Minor criteria a, b and c

  * Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of ≥ 1 g/dL and/or urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours.
  * Non-secretors must have measurable protein by Freelite or measurable disease such as plasmacytoma to be eligible.
  * Has asymptomatic disease, i.e., does not have hypercalcemia, renal insufficiency, anemia or bone lesions.
  * Karnofsky performance status ≥ 80 (See Appendix B)
  * Is infertile (i.e. surgically sterile or 12 months post-menopausal) or is practicing an adequate form of contraception, as judged by the investigator (i.e., birth control pills, double barrier method, abstinence, etc.)
  * Age 18 years or older
  * Has given voluntary written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior treatment for myeloma (symptomatic or asymptomatic).
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
* Plasma cell leukemia
* Patients with a history of thyroid problems.
* Receiving steroids > the equivalent of 10 mg prednisone daily for other medical conditions, e.g., asthma, systemic lupus erythematosis, rheumatoid arthritis
* Infection not controlled by antibiotics
* Human Immunodeficiency Virus (HIV) infection. Patients should provide consent for HIV testing according to the institution's standard practice
* Known active hepatitis B or C
* New York Hospital Association (NYHA) Class III or IV heart failure or EKG evidence of acute ischemic disease
* Second malignancy requiring treatment in last 3 years
* Other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Positive pregnancy test in women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabha Mazumder, MD, Principal Investigator — NYU School of Medicine, Clinical Cancer Center
Locations (1):
- New York University School of Medicine, Clinical Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2011 to October 2012, 20 patients were enrolled to the study from Perlmutter Cancer Center at NYU Lagone Medical Center.
Groups:
- Sea Cucumber Extract (TBL 12): TBL12 is administered orally at a dose of 2 units (of 20 mL each) twice a day, in 4-week cycles, until disease progression or there is sign of disease progression.
Period: Overall Study
Arm/Group | Sea Cucumber Extract (TBL 12)
Started | 20
Completed | 15
Not Completed | 5
Not completed — patient choice or noncompliance | 5

BASELINE CHARACTERISTICS:
Groups:
- Sea Cucumber Extract (TBL 12): TBL12 is administered orally at a dose of 2 units (of 20 mL each) twice a day, in 4-week cycles, until disease progression or there is sign of disease progression.
  TBL-12
Arm/Group | Sea Cucumber Extract (TBL 12)
Number analyzed (Participants) | 20
Age, Customized [Number; unit: participants]
  35-44 years | 1
  45-53 years | 2
  54-63 years | 9
  64-73 years | 5
  74-83 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Duration of Response (All Treated Patients)
Description: Response [complete response (CR), partial response (PR), and stable disease (SD)] was assessed after approximately 2 months, 6 months and then every 4 months, until progression of disease. Response and progression of disease evaluation is based on the criteria reported by Blade, et al. (1998).
Time Frame: up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Sea Cucumber Extract (TBL 12)
Number analyzed (Participants) | 20
months | 19.7 [2.0 to 31.0]

2. Secondary Outcome: Percentage of Patients Who Have Responded to TBL12
Description: Response to TBL12 is defined as SD or better after 2 cycles of TBL12. The evaluation of SD, PR, or CR is based on the report by Blade et al. (1998)
Time Frame: 2 months
Population: all patients
Measure: Number; unit: percentage of participants
Arm/Group | Sea Cucumber Extract (TBL 12)
Number analyzed (Participants) | 20
percentage of participants | 100

3. Primary Outcome: Duration of Response (Excluding Patient Choice and Non-compliance)
Description: as for outcome 1
Time Frame: up to 3 years
Population: All patients or the patients excluding personal choice or non-compliance
Measure: Median (Full Range); unit: months
Arm/Group | Sea Cucumber Extract (TBL 12)
Number analyzed (Participants) | 15
months | 21.0 [8.5 to 31.0]

ADVERSE EVENTS:
Time Frame: up to one year
Description: All adverse events regardless of attribution are reported here.
Arm/Group | Sea Cucumber Extract (TBL 12)
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sea Cucumber Extract (TBL 12) (N=20)
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection with Grade 3 or 4 neutrophils: Skin (cellulites) (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sea Cucumber Extract (TBL 12) (N=20)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Rash: acne/acneiform: (Skin and subcutaneous tissue disorders) | 3
Mood alteration: Agitation (Psychiatric disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Mood alteration: Anxiety (Psychiatric disorders) | 1
Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Arthritis (non-septic): (Musculoskeletal and connective tissue disorders) | 2
Pain: Back (Musculoskeletal and connective tissue disorders) | 9
Infection with normal ANC or Grade 1 or 2 neutrophils: Bladder (urinary) (Infections and infestations) | 2
Creatinine (Metabolism and nutrition disorders) | 2
Pain: Bone (Musculoskeletal and connective tissue disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Bronchus (Infections and infestations) | 3
Pain: Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 1
Perforation, GI: Colon (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Mood alteration: Depression (Psychiatric disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8
Flatulence (Gastrointestinal disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1
Pain: Intestine (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Pain: Head/headache (Nervous system disorders) | 6
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Flu-like syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Insomnia (Psychiatric disorders) | 1
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytes (total WBC) (Investigations) | 2
Memory impairment (Nervous system disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils: Mucosa (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 5
Pain: Neck (Musculoskeletal and connective tissue disorders) | 3
Pain: Neuralgia/peripheral nerve (Nervous system disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 14
Pain: Pelvis (Reproductive system and breast disorders) | 1
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 3
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Lung (pneumonia) (Infections and infestations) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Fever (in the absence of neutropenia) (General disorders) | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1
Rigors/chills (General disorders) | 2
Seroma (Musculoskeletal and connective tissue disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Sinus (Infections and infestations) | 2
Pain: Stomach (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic): Oral cavity (Gastrointestinal disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 1
Urinary retention (including neurogenic bladder): (Renal and urinary disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Urinary tract NOS (Infections and infestations) | 2
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Vagina (Infections and infestations) | 1
Vision-blurred vision (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (General disorders) | 1
Pain: Buttock (Musculoskeletal and connective tissue disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Upper airway NOS (Infections and infestations) | 10
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Stomach (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils: Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Allergic reaction/ hypersensitivity (Immune system disorders) | 5
Cardiac General - Other: heart flutter (Cardiac disorders) | 1
Infection - Other: staph infection (skin) (Infections and infestations) | 1
Metabolic/Laboratory - Other: elevated BUN (Metabolism and nutrition disorders) | 1
Dry Eyes (Eye disorders) | 1
Pain NOS (General disorders) | 3
Nasal Cavity/Paranasal Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1
Infection with unknown ANC: Sinus (Infections and infestations) | 1
Infection with unknown ANC: Vagina (Infections and infestations) | 1
Edema: limb (General disorders) | 2
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 2
Infection, other: upper respiratory infection (Infections and infestations) | 1
Infection, other: abdominal infection (Infections and infestations) | 1
Dermatology/skin, other: finger splinter (Skin and subcutaneous tissue disorders) | 1
Allergy/Immunology, other: autoimmune disorder (Immune system disorders) | 1
Pain, other: hip (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes